CLINICAL TRIAL: NCT06120179
Title: Recombinant tPA by Endovascular Pulse Administration for the Treatment of Submassive Pulmonary Embolism Using Pharmaco-mechanical Catheter Directed Thrombolysis for the redUction of Thrombus burdEn
Brief Title: The RESCUE II Study. The Bashir™ Endovascular Catheter (BEC),
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: The RESCUE II Study
Record Dates: First submitted 2023-10-26; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Acute Submassive Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, multi-center study. The Bashir™ Endovascular Catheter (BEC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Patients who present with PE (Experimental): The Bashir™ Endovascular Catheter (BEC) is a device intended for the localized infusion of therapeutic agents into the pulmonary artery and peripheral vasculature. Two sizes of BECs will be used in this study
  Interventions: Device: The Bashir™ Endovascular Catheter (BEC

INTERVENTIONS:
Device: The Bashir™ Endovascular Catheter (BEC — To demonstrate the efficacy and safety of the Bashir™ Endovascular Catheter for the administration of pharmaco-mechanical catheter directed therapy using pulse spray of r-tPA for the treatment of acute submassive pulmonary embolism.

SUMMARY:
To demonstrate the efficacy and safety of the Bashir™ Endovascular Catheter for the administration of pharmaco-mechanical catheter directed therapy using pulse spray of r-tPA for the treatment of acute submassive pulmonary embolism

DETAILED DESCRIPTION:
Study Objective To demonstrate the efficacy and safety of the Bashir™ and Bashir™ S-B Endovascular Catheters for the administration of pharmaco- mechanical catheter directed therapy in a pulse spray mode using low dose r-tPA for the treatment of acute submassive pulmonary embolism. Endpoints Primary Efficacy Endpoint Reduction in RV/LV diameter ratio as measured by CTA within 48 hours after the completion of r-tPA treatment.

Primary Safety Endpoint Major bleeding, as defined by International Society of Thrombosis and Hemostasis (ISTH), within 72 hours of initiation of r- tPA infusion. ISTH major bleeding in non-surgical patients is defined as having a symptomatic presentation and:

a. Fatal bleeding; and/or b. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra- articular or pericardial, or intramuscular with compartment syndrome; and/or c. Bleeding causing a fall in hemoglobin level of 2.0g/dL (1.24mmol/L) or more or leading to transfusion of two or more units of whole blood or red cells. Secondary Endpoints

1. Refined Modified Miller Score as measured on CTA within 48 hours after the completion of the r-tPA infusion compared to baseline as measured by core lab. 25
2. All-cause mortality at hospital discharge through 30-day follow-up.
3. SAEs through 30-day follow-up.
4. AEs through 30-day follow-up.
5. UADEs through 30-day follow-up.
6. Recurrent PE through 30-day follow-up.
7. Clinically Relevant Non-Major bleeding: Any sign or symptom of hemorrhage (e.g. more bleeding than would be expected for a clinical circumstance, including bleeding found by imaging alone) that does not fit the criteria for the ISTH definition of major bleeding but does meet at least one of the following criteria:

   1. Requiring medical intervention by a healthcare professional.
   2. Leading to hospitalization or increased level of care.
   3. Prompting a face to face (i.e., not just a telephone or electronic communication) evaluation.
8. Technical procedural complications.
9. Systolic PA pressure measured at completion of pulse sprays and after BEC(s) removal and compared to baseline.
10. Cardiac output (CO by Modified Fick calculation) and cardiac index (CI) following completion of the r-tPA pulse sprays compared to the baseline. Please refer to Terms and Definitions section for the Modified Fick calculation to be done in the IR suite / cath lab at baseline and after BEC removal).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  1. Willing and able to provide informed consent;
  2. Age 18 to ≤ 75 years of age;
  3. PE symptom duration ≤ 14 days.
  4. Filling defect in at least one main or lobar pulmonary artery as determined by CTA;
  5. RV/LV diameter ratio ≥ 0.9 by CTA as determined by the investigative site;
  6. Willing and able to comply with all study procedures and follow-up

Exclusion Criteria:

1. CVA or TIA within one (1) year;
2. Head trauma, active intracranial, or intraspinal disease ≤ one (1) year prior to inclusion in the study;
3. Active bleeding from a major organ within one (1) month prior to inclusion in the study;
4. Intracranial condition(s) that may increase the risk of bleeding (e.g., neoplasms, arteriovenous malformations, or aneurysms);
5. Patients with bleeding diatheses;
6. Hematocrit < 30%;
7. Platelets < 100,000/μL;
8. INR > 1.5 if currently on warfarin (Coumadin®);
9. aPTT > 50 seconds in the absence of anticoagulants;
10. Major surgery ≤ 14 days prior to inclusion in the study;
11. Serum creatinine > 2.0mg/dL;
12. Clinician deems high-risk for catastrophic bleeding;
13. History of heparin-induced thrombocytopenia (HIT Syndrome);
14. Pregnancy;
15. SBP < 90 mmHg > 15 minutes within two (2) hours prior to BEC procedure and is not resolved with IV fluids;
16. Any vasopressor support;
17. Cardiac arrest (including pulseless electrical activity and asystole) requiring active cardiopulmonary resuscitation (CPR) during this hospitalization at treating institution and/or referring institution;
18. Evidence of irreversible neurological compromise;
19. Life expectancy < one (1) year;
20. Use of thrombolytics or glycoprotein IIb/IIIa inhibitor within 3 days prior to inclusion in the study;
21. Profound bradycardia requiring a temporary pacemaker and/or inotropic support;
22. Absolute contraindication to anticoagulation;
23. Uncontrolled hypertension defined as SBP > 175mmHg and / or DBP > 110mmHg with pharmacotherapy within two (2) hours prior to inclusion in the study;
24. Currently participating in another study;
25. In the opinion of the investigator, the subject is not a suitable candidate for the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in RV/LV diameter ratio as measured by contrast enhanced chest CT from baseline within 48 ± 6 hours of initiation of treatment. chest CT (CTA) within 48 hours after the completion of r-tPA treatment | Through 30 day follow-up
  Reduction in RV/LV diameter ratio as measured by contrast enhanced chest CT (CTA) within 48 hours after the completion of r-tPA treatment
Primary Safety Endpoint, major bleeding, as defined by International Society of Thrombosis and Hemostasis (ISTH), within 72 hours of initiation of rtPA infusion. ISTH major bleeding in non-surgical patients is defined as having a symptomatic presentation | 72 hours
  Major bleeding, as defined by International Society of Thrombosis and Hemostasis (ISTH), within 72 hours of initiation of rtPA infusion. ISTH major bleeding in non-surgical patients is defined as having a symptomatic presentation and:
  1. Fatal bleeding; and/or
  2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome; and/or Bleeding causing a fall in hemoglobin level of 2.0g/dL (1.24mmol/L) or more or leading to transfusion of two or more units of whole blood or red cells

SECONDARY OUTCOMES:
Refined Modified Miller Score | Within 48 hours of completion of r-TPA
  Refined Modified Miller Score as measured on CTA within 48 hours after the completion of the r-tPA infusion compared to baseline as measured by core lab
All-cause mortality | 30 DAYS
  All-cause mortality at hospital discharge through 30-day follow-up.
Serious adverse events | 30 days
  Serious adverse events through 30-day follow-up
Adverse events | 30 days
  Adverse events through 30-day follow-up
Unanticipated adverse device events | 30 days
  Unanticipated adverse device events through 30-day follow-up
Recurrent pulmonary embolism through 30-day follow-up. | 30 days
  Recurrent pulmonary embolism through 30-day follow-up.
Clinically relevant non-major bleeding | 30 days
  Any sign or symptom of hemorrhage (e.g. more bleeding than would be expected for a clinical circumstance, including bleeding found by imaging alone) that does not fit the criteria for the ISTH definition of major bleeding but does meet at least one of the following criteria:
  1. Requiring medical intervention by a healthcare professional.
  2. Leading to hospitalization or increased level of care.
  3. Prompting a face to face (i.e., not just a telephone or electronic communication) evaluation
Technical procedural complications. | 1 day
  Technical procedural complications.
Systolic PA pressure | Once r-tPA pulse sprays are given continue therapeutic anticoagulation with full does heparin or LMWH with sheaths sutured in place
  Systolic PA pressure measured at completion of pulse sprays and after BEC(s) removal and compared to baseline
Cardiac output (CO by Modified Fick calculation) and cardiac index (CI) following completion of the r-tPA pulse | End of procedure
  Cardiac Index: Hemodynamic parameter that relates the cardiac output (CO) from right or left ventricle in one minute to body surface area (BSA), thus relating heart performance to the size of the individual. The unit of measurement is liters per minute per square meter (L/min/m2 ). CI = CO/BSA

CONTACTS AND LOCATIONS:
Overall Officials: Parth Rali, MD, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No